CLINICAL TRIAL: NCT03377530
Title: Contamination of Bacillus Species Sepsis.
Acronym: BACILLUS
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD1715
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Bacillus Cereus Infection
Keywords: Bacillus Cereus; Premature neonates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Premature neonates infected with bacillus Species: The investigators studied retrospectively eleven cases of these infections in our NICU and reviewed series and report cases in literature.
  Interventions: Diagnostic Test: Ways to prevent these infections.

INTERVENTIONS:
Diagnostic Test: Ways to prevent these infections. — The purpose of this database is to describe the pathogenicity of this germ, the incriminated modes of contamination.
  The collaborators studied the factors of poor prognosis and propose ways to prevent these infections.

SUMMARY:
Bacillus species are ubiquitous gram-positive spore-forming organisms. They rarely cause disease in the immunocompetent and are more frequently isolated as a culture contaminant. However, Bacillus Species can cause severe systemic infections in immunocompromised patients including preterm infants.

The purpose of this study is to identify the risk factors of these infections.

DETAILED DESCRIPTION:
Non-anthrax Bacillus Species bacteria can be responsible for food poisoning and local infections. Rarely, they lead to severe infections like blood stream infections and meningitis especially in immunocompromised patients like preterm infants.

Bacillus Cereus is the most common members of the genus Bacillus. Only few reports studied these systemic infections in premature neonates. In order to identify the risk factors for severe Bacillus Species infections, we studied retrospectively eleven cases of these infections in our NICU and reviewed series and report cases in literature.

ELIGIBILITY:
Inclusion Criteria:

* cases of Bacillus Species sepsis
* cases of Bacillus species meningitis
* with significant change in clinical status
* Bacillus Species is the only organism isolated

Exclusion Criteria:

* Bacillus Species isolated with other organisms and Bacillus Species without clinical change were considered to be contaminants

Max Age: 28 Days | Sex: All
Age Groups: Child
Study Population: Newborns infected with Bacillus Species.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Severe infection rate due to Bacillus Sp germ | Through study completion, an average of 1 year.
  The purpose of this database is to mesure the pathogenicity of this germ based on the severe infection rate

SECONDARY OUTCOMES:
To collecte the incriminated modes of contamination. | Through study completion, an average of 1 year.
  The purpose of this database is to describe the incriminated modes of contamination.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Amine YANGUI, Principal Investigator — Hôpital NOVO

IPD SHARING:
Plan to Share IPD: No